CLINICAL TRIAL: NCT02711332
Title: Investigating the Influence of Haemolysis on the Potassium Concentration After Capillary Blood Sampling
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Collaborators: Joanneum Research Forschungsgesellschaft mbH (Other)
Responsible Party: Sponsor
Other Study IDs: K@Home_1
Record Dates: First submitted 2015-11-24; First posted 2016-03-17 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Hemolysis
MeSH Terms: conditions — Hemolysis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Degree of Haemolysis: Each subject will have four capillary blood sampling on different fingers. A reference venous blood sampling will be conducted.
  Interventions: Other: capillary blood sampling; Other: venous blood sampling

INTERVENTIONS:
Other: capillary blood sampling — Each subject will have four capillary blood collections on different fingers. A reference venous blood collection will be conducted.
  Other Names: capillary blood sampling on fingertips
Other: venous blood sampling — Each subject will have four capillary blood collections on different fingers. A reference venous blood collection will be conducted.
  Other Names: blood sampling

SUMMARY:
This is an open, single-centre trial investigating the impact of haemolysis after capillary blood collection to the measured potassium concentration in Plasma healthy subjects. Each subject will have four capillary blood collections on different fingers. Two on the right and two on the left hand. Additionally as a reference a venous blood collection will be conducted.

DETAILED DESCRIPTION:
K@Home_1 a working package of the FFG project "K@Home - potassium home monitoring for patients with heart- and kidney insufficiency". In the project K@Home a potassium measuring system serveable by the patients even of the home monitoring should be developed.

Aim from K@Home is to allow an everyday home monitoring of the potassium value by the development of potassium-test stripe, like with the diabetes patients who supervise their blood sugar level by measurements with glucose-test stripe from a drop of capillary blood from the finger berry and with it the emergencies and hospital admissions to reduce or to prevent. It is fact that haemolysis has a strong influence on the measured potassium concentration. It is likely that by using capillary blood a haemolysis appears and therefore distorted potassium concentrations are measured.

In the study K@Home_1 it is a matter of evaluating, how high the degree of the haemolysis in capillary blood is, and in this fact to what extent leads to wrong potassium values. The results from this study will be a basic component for the sensor development.

After clarification the approval the Informed Consent is signed and the inclusion as well as exclusion criteria (incl. demography, concomitant medication and medical history) or vital parameters (blood pressure, pulse, size, weight), are raised. An urine-pregnancy test is also carried out for the exclusion of a pregnancy in women capable of bearing children. It is not necessary that the subjects seem sober on the study day.

With 22 healthy subjects capillary and venous blood is taken within the scope of one single study round. Blood is taken from the test persons by trained specialist staff of two fingertips of each hand (a total of four fingertips). The capillary blood sampling occurs in 200 µ l Lithium-Heparin Sarsted Microvettes and in each case the first drop of blood is rejected. To guarantee a light blood decrease without strong mechanical pressure, the hands are warmed up before the capillary sampling required with the help of an electric blanket or by warm water roughly on room temperature.

In addition 15 ml blood from the vein of a forearm is taken.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Healthy
* Signed informed consent before any trial-related activities

Exclusion Criteria:

* Severe acute and/or chronic diseases
* Mental incapacity, unwillingness of language barriers precluding adequate understanding or cooperation
* Pregnancy or breastfeeding
* Any disease or condition which the investigator or treating physician feels would interfere with the trial or the safety of the subject

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Communtiy Sample
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2015-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Measured potassium concentration in capillary blood tests compared to venous blood tests. | 1 hour

SECONDARY OUTCOMES:
Correlation from fHb and potassium | 1 hour
Degree of haemolysis in capillary blood tests compared to venous blood tests. | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Julia Mader, Prof.Dr., Principal Investigator — Medical University of Graz